CLINICAL TRIAL: NCT01731795
Title: A Comparative, Randomised Controlled Trial for Evaluating the Efficacy of Dexamethasone in the Treatment of Patients With Acute Respiratory Distress Syndrome
Brief Title: Efficacy Study of Dexamethasone to Treat the Acute Respiratory Distress Syndrome
Acronym: DEXA-ARDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Fundación Mutua Madrileña (Other); Asociación Científica Pulmón y Ventilación Mecánica (Other)
Responsible Party: Principal Investigator, Jesus Villar, Director of Research, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-000775-17
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome, mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No dexamethasone (No Intervention): Patients will be treated with conventional treatment
- Dexamethasone (Active Comparator): Conventional treatment plus dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone (20 mg/iv/daily/from Day 1 of randomization during 5 days, followed by 10 mg/iv/daily/ from Day 6 to 10 of randomization)
  Other Names: Dexamethasone Indukern
  Arms: Dexamethasone

SUMMARY:
BACKGROUND: Currently, there is no proven pharmacologic treatment for patients with the acute respiratory distress syndrome (ARDS). Great interest remains in the use of corticosteroids for the salvage of patients with severe acute lung injury in the early phase of their disease process, a situation that that has not been evaluated in most published trials. Dexamethasone has never been evaluated in ARDS in a randomized controlled fashion.

HYPOTHESIS AND OBJECTIVES: The investigators hypothesize that adjunctive treatment with intravenous dexamethasone of patients with established ARDS might change the pulmonary and systemic inflammatory response and thereby will increase the number of ventilator-free days and will decrease the extremely high overall mortality. Our goal is to examine the effects of dexamethasone on length of duration of mechanical ventilation (assessed by number of ventilator-free days) and on mortality, in patients admitted into a network of Spanish intensive care units (ICUs) who still meet ARDS criteria at 24 hours after ARDS onset.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is an inflammatory disease process of the lungs as a response to both direct and indirect insults, characterized clinically by severe hypoxemia, reduced lung compliance, and bilateral radiographic infiltrates. ARDS is caused by an insult to the alveolar-capillary membrane that results in increased permeability and subsequent interstitial and alveolar edema. The mechanisms by which a wide variety of insults can lead to this syndrome are not clear. It is useful to think of the pathogenesis of ARDS as a result of two different pathways: a direct insult on lung cells and an indirect insult as a result of an acute systemic inflammatory response.

Like any form of inflammation, acute lung injury during ARDS represents a complex process in which multiple cellular signalling pathways can propagate or inhibit lung injury. Death has traditionally been attributed to the underlying disease, the presence of sepsis and the failure of vital organ systems other than the lung. The association of ARDS with multiple system organ dysfunctions is not inevitable, but it certainly is common. It is postulated that local injury to the lungs (pneumonia, trauma, aspiration, gas inhalation) could set up a secondary diffuse inflammatory response resulting in damage to other organs.

Although much has evolved in our understanding of its pathogenesis and factors affecting patient outcome, still there is no specific pharmacologic treatment for ARDS. Despite advances in supportive measures and antibiotics, ARDS has a mortality rate of about 40-50% in most series and it is associated with significant health care costs. Patients with ARDS invariably require endotracheal intubation and mechanical ventilation (MV) to decrease the work of breathing and to improve oxygen transport. To date the only proven, widely accepted method of MV for ARDS is what is called "lung protective ventilation" using a low tidal volume strategy plus positive end-expiratory pressure (PEEP).

Corticoids seemed to be an ideal therapy for the acute lung injury in ARDS, given their potent anti-inflammatory and antifibrotic properties. They switch off genes that encode pro-inflammatory cytokines and switch on genes that encode anti-inflammatory cytokines. It has been reported that low doses of corticosteroids prevent an extended cytokine response and might accelerate the resolution of pulmonary and systemic inflammation in pneumonia.

Dexamethasone has never been evaluated in ARDS in a randomized controlled fashion. However, dexametasone has potent anti-inflammatory effects and weak mineralocorticoid effects compared with other corticosteroids. Dexamethasone has a long-lasting effect, allowing for a once-a-day regimen. Whether addition of dexamethasone to conventional supportive treatment benefits ARDS patients is unknown, it has been used in patients with sepsis, septic shock, pneumonia, trauma, and meningitis, all of them causes of ARDS.

The investigators justify the need of our study based on the positive results of two recent clinical trials: (i) Meijvis et al (Lancet 2011) showed that dexamethasone (5 mg/day) for 4 days was able to reduce length of hospital stay in 304 patients with bacterial pneumonia when added to the conventional treatment; (ii) Azoulay et al (Eur Respir J 2011) showed that dexamethasone (10 mg/6h), when added to chemotherapy and conventional ICU management, caused less respiratory deterioration and lower ICU mortality in 40 patients with acute lung injury resulting from leukaemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients must have acute onset of ARDS, as defined by the American-European Consensus Conference (AECC) criteria for ARDS: (i) having an initiating clinical condition (pneumonia, aspiration, inhalation injury, sepsis, trauma, acute pancreatitis, etc.; (ii) bilateral infiltrates on frontal chest radiograph; (iii) absence of left atrial hypertension, a pulmonary capillary wedge pressure (PCWP) less than 18 mm Hg, or no clinical signs of left heart failure; (iv) severe hypoxemia (a PaO2/FIO2 <200 mm Hg, regardless of FIO2 or positive end-expiratory pressure (PEEP)
* Be intubated and mechanically ventilated
* Have provided signed written informed consent from the patient or the patient's personal legal representative

Exclusion Criteria:

* Be a woman known to be pregnant or lactating
* Take part in another experimental treatment protocol (simultaneously)
* Brain death
* Terminal-stage cancer or other terminal disease
* Having do-not-resuscitate orders
* Being immune-compromised
* Receiving corticosteroids or immunosuppressive drugs
* Patients in whom more than 24 hours had elapsed after initially meeting the AECC ARDS criteria before consent and results of initial standard ventilator settings could be obtained.
* Have severe chronic obstructive pulmonary disease (COPD)
* Have congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Ventilator free-days | 28 days
  Number of ventilator free-days (VFDs) at Day 28 (defined as days alive and free from mechanical ventilation at day 28 after intubation. For subjects ventilated ≥28 days and for subjects who die, VFD is 0.

SECONDARY OUTCOMES:
Mortality | 60 days
  All-cause mortality at Day 60 after enrolment.

OTHER OUTCOMES:
organ failure | ICU discharge
  Number of extrapulmonary organ system failures

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Research Unit, Hospital Universitario Dr. Negrín, Las Palmas, Spain
Locations (2):
- Spain (2):
  - Hospital Universitario Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Clinico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Derived] Sweeney RM, McAuley DF. Prolonged glucocorticoid treatment in acute respiratory distress syndrome - Authors' reply. Lancet. 2017 Apr 15;389(10078):1516-1517. doi: 10.1016/S0140-6736(17)30953-4. No abstract available. PMID 28422025
- [Derived] Villar J, Belda J, Anon JM, Blanco J, Perez-Mendez L, Ferrando C, Martinez D, Soler JA, Ambros A, Munoz T, Rivas R, Corpas R, Diaz-Dominguez FJ, Soro M, Garcia-Bello MA, Fernandez RL, Kacmarek RM; DEXA-ARDS Network. Evaluating the efficacy of dexamethasone in the treatment of patients with persistent acute respiratory distress syndrome: study protocol for a randomized controlled trial. Trials. 2016 Jul 22;17:342. doi: 10.1186/s13063-016-1456-4. PMID 27449641